CLINICAL TRIAL: NCT00386048
Title: Home-based Pain Management Protocol for Children With Sickle Cell Disease
Brief Title: Pain Management Protocol for Pediatric Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: SCD pain management protocol
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Sickle Cell Disease
Keywords: Cognitive Behavioral Therapy; Pediatric Sickle Cell Disease; Pain Management
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard of Care Observation Group: This group is randomized to continue their current medical management strategies for pain as recommended/prescribed by health care providers. Primary and secondary outcomes are collected at the same time intervals as the biopsychosocial intervention group.
- Biopsychosocial Intervention Group: This group continues all standard of care procedures for managing pain and adds to this additional cognitive-behavioral treatment (CBT) strategies for managing pain. The intervention explicitly frames the CBT strategies as added, complimentary pain management methods to add to the standard of care treatment.
  Interventions: Behavioral: Brief Cognitive-Behavioral Pain Management Training

INTERVENTIONS:
Behavioral: Brief Cognitive-Behavioral Pain Management Training — Participants complete a manualized, single session of training which includes: (A) education about the causes of sickle cell pain, (B) education about how the nervous system processes pain signals, and (C) explanations of how one can use cognitive and behavioral treatment (CBT) strategies to decrease the extent of pain experienced (all based on how the nervous system processes pain). Four specific CBT skills are taught and practiced by the participant (Progressive muscle relaxation, Controlled Deep Breathing, Imagery, and Distraction). The protocol explicitly emphasizes the use of CBT as a complimentary pain management tool to use in addition to the standard of care methods.
  Groups: Biopsychosocial Intervention Group

SUMMARY:
Sickle cell disease (SCD) is a devastating chronic health condition that primarily affects African-Americans. Painful episodes are the most frequent form of morbidity in SCD and the most frequent reason for hospitalization. Cognitive-behavioral interventions for pain management have shown efficacy for improving coping abilities, reducing the amount of medication needed to manage pain, and improving daily functioning during painful episodes. However, difficulties with disseminating and implementing cognitive-behavioral treatments have resulted in almost no use of these techniques in pediatric settings. In South Carolina these difficulties are compounded by social and geographical factors that pose particular challenges. A major issue with implementing quality pain management protocols is the difficulty with providing adequate practice and monitoring of the use of the techniques, particularly given the rural population in South Carolina and transportation difficulties for economically disadvantaged families. Due to a history of under-treating pain in SCD it is also critical that psychological and medical treatments are presented in an integrated manner so that these approaches are viewed as complimentary, not mutually exclusive, approaches to pain management. Finally, we believe the same implementation issues for improving the use of behavioral coping skills are also important for improving adherence to medication protocols for appropriate home-based pain management.

The purpose of this proposal is to develop, implement, and evaluate a pain management protocol that uses portable electronic devices and other technologies to increase the practice of psychosocial pain management techniques, improve adherence to the overall biopsychosocial pain management protocol, and improve the clinician's ability to track progress with fewer office visits. In addition to addressing important dissemination issues, by embedding methods to assess for adherence into the technology it will be possible to continuously evaluate and modify protocol efficacy, resulting in a product that is effective, empirically sound, and flexible. Participants will be randomly assigned to the intervention or waitlist control condition. Those on the waitlist condition will receive the same study procedures after a 2 month wait periods. We anticipate that the intervention will result in better pain management and less impairment in the participants.

DETAILED DESCRIPTION:
"Home-Based Pain Management Protocol for Children with Sickle Cell Disease"

BACKGROUND: Sickle cell disease (SCD) is a devastating chronic health condition that primarily affects African-Americans. Painful episodes are the most frequent form of morbidity in SCD and the most frequent reason for hospitalization. Cognitive-behavioral interventions for pain management have shown efficacy for improving coping abilities, reducing the amount of medication needed to manage pain, and improving daily functioning during painful episodes. However, difficulties with disseminating and implementing cognitive-behavioral treatments have resulted in almost no use of these techniques in pediatric settings. In South Carolina these difficulties are compounded by social and geographical factors that pose particular challenges. A major issue with implementing quality pain management protocols is the difficulty with providing adequate practice and monitoring of the use of the techniques, particularly given the rural population in South Carolina and transportation difficulties for economically disadvantaged families. Due to a history of under-treating pain in SCD it is also critical that psychological and medical treatments are presented in an integrated manner so that these approaches are viewed as complimentary, not mutually exclusive, approaches to pain management. Finally, we believe the same implementation issues for improving the use of behavioral coping skills are also important for improving adherence to medication protocols for appropriate home-based pain management.

PURPOSE: The purpose of this research is to implement and evaluate a pain management protocol that uses portable electronic devices (PDA) and other technologies to increase the practice of psychosocial pain management techniques, improve adherence to the overall biopsychosocial pain management protocol, and improve the clinician's ability to track progress with fewer office visits. In addition to addressing important dissemination issues, by embedding methods to assess for adherence into the technology it will be possible to continuously evaluate and modify protocol efficacy, resulting in a product that is effective, empirically sound, and flexible.

STUDY PROCEDURES:

Recruitment and Assignment to Study Conditions. Families will be approached as part of their routine psychosocial screenings currently conducted at the Children's Cancer and Blood Disorder Center. Parental informed consent and child assent will be obtained from families who meet inclusion criteria and agree to participate. Next, participants will be randomly assigned to waitlist control or intervention groups through the use of a random assignment procedure. The researcher will explain details of the participation incentive system to the families at this time, including the number of coupons assigned for each phase of study completion and how to redeem coupons for toys and gift cards. All participants (waitlist control group and intervention group) will complete the initial measures: Background Information Questionnaire ; Structured Pain History Interview - Parent and Child Forms; Coping Strategies Questionnaire (CSQ); Pediatric Quality of Life Inventory (PEDS-QL); Pediatric Pain Questionnaire (PPQ); Child Health Locus of Control during the initial meeting and the second set of measures (CSQ, PEDS-QL and PPQ) 4 weeks after the initial meeting.

Cognitive-Behavioral Training. Following completion of the intake measures, families in the intervention condition will be provided education on pain medication use and explanation of active versus passive methods of coping with pain and the cognitive-behavior techniques will be introduced (Progressive Muscle Relaxation, Deep Breathing, Guided imagery and Distraction). These techniques will be tailored to the child's preferences and recorded onto the PDA.

Next, the researcher will review with the family the pain flow chart, how to complete the Daily Pain and Activity Diary (DPAD), and use the PDA and Pain Management software. Participants and their parents will be provided with detailed instructions regarding care of PDA, who to contact if device is broken or lost, policy on continued participation if device is lost, and a padded addressed stamped envelope to return the PDA should it require attention. Three days after the initial visit families will be contacted to answer questions and ensure implementation of skills.

Families will also receive a weekly telephone contact at a pre-arranged time to address any difficulties with protocol implementation. Pain diaries and frequency of skills practice will be electronically downloaded approximately every three days using wireless synchronization built into the PDA devices. One month following the initial session, all participants (waitlist and intervention groups) will complete the PPQ, PEDS-QL and CSQ outcome measures. Two months after the initial session, intervention participants will complete outcome measures, including PPQ, PEDS-QL, CSQ and Protocol Evaluation Form (PEF). Six months after the initial session, intervention participants will complete the follow-up measures, including child report on the CSQ, and parent and child report on the PPQ and PEDS-QL. At this time the participant's school will be contacted to obtain school attendance records so as to document absences due to illness over the previous year and participants medical records will be reviewed to examine patient's disease severity over the course of their study participation time and their lives (Medical Record Review Form). Participants in the waitlist control group will start participation in the intervention at the two month point, and follow the procedures outlined above for the intervention condition.

Concurrent Validity Study Procedures. Assessment of pain experience will be obtained for study participants undergoing routine venipuncture as part of their clinic visit co-occurring with study entry and study completion. Observational, physiological response, parent-report, and self-report of pain experience will be obtained to provide convergent validity for measures of pain report. A brief measure of medical coping style, the Child Approach-Avoidance Rating Scale (CAARS; Appendix J) will be included to assess for shifts in coping strategies employed by the participant during painful procedures. Participants and parents will report on child pain experience before, during, and after the routine venipuncture that is part of their clinic visit on the day of initial contact. Participant response to routine venipuncture will also be captured via video recording to allow for an in-depth analysis of observable pain behaviors. Pre-procedural heart rate will be taken at three intervals: when the patient is first seen for the clinic visit, immediately prior to the venipuncture, and immediately following the venipuncture. Additionally, small extra vial of blood will be obtained (5mL) to measure the participant's level of endothelin-1, a biological marker of pain. This extra vial of blood will not require an additional needle stick. Finally, the medical records of all participants will be reviewed to obtain information about disease course.

SUBJECT POPULATION:

Participants will include up to 50 children and adolescents with SCD ranging between the ages of 8 to 18 years of age and their primary caregivers. Participants will be recruited from the Children's Cancer and Blood Disorder Center at Palmetto Health and four DHEC Children's Rehabilitative Services sites (Orangeburg, Columbia, Florence and Sumter). Reviews of behavioral interventions for rheumatoid arthritis or chronic low back pain have indicated typical treatment effect sizes for pain experience and coping of d = 0.46 or greater (Astin et al., 2002; van Tulder et al., 2001). Using this value as a basis for computing study power (with an alpha level of .05) the study has an expected power of .80 with a sample size of 50 participants.

Inclusion/Exclusion criteria:

Inclusion criteria mandate that the families selected demonstrate adherence with standard SCD treatment as indicated by reliable attendance to clinic visits, and chart notes demonstrating adherence to prescribed medical care (e.g., follow-through with required specialist visits and appointments for diagnostic procedures). Participants must have had at least 1 major pain episode or 3 minor pain episodes in the previous 6 months that resulted in functional impairment, such as reduced school attendance. Finally, individuals with developmental disabilities such as mental retardation, autism, and Down syndrome, severe cognitive limitations following stroke, or diagnoses of severe psychopathology will be excluded from participation as these disorders have the potential to confound the findings.

CONFIDENTIALITY: To minimize threats to confidentiality, only investigators will have access to participant data. For data management purposes and confidentiality, subjects will be given a unique identifier to use when recording data and electronically transmissions of data. This arrangement minimizes risk to loss of patient confidentiality. All study staff, including research assistants who may enter data, will be required to complete and pass the University of South Carolina Human Subjects on-line tutorial prior to commencing their work on this research project. All data will be stored in a locked file cabinet in the investigators office at Palmetto Health.

EXPECTED RESULTS AND IMPLICATIONS: We anticipate that the intervention will result in better pain management and less impairment in the participants. These data will be used to seek funding for a larger-scale study and in the development of interventions to decrease the impact of pain on the lives of individuals with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria mandate that the families selected demonstrate adherence with standard SCD treatment as indicated by reliable attendance to clinic visits, and chart notes demonstrating adherence to prescribed medical care (e.g., follow-through with required specialist visits and appointments for diagnostic procedures). Participants must have had at least 1 major pain episode or 3 minor pain episodes in the previous 6 months that resulted in functional impairment, such as reduced school attendance.

Exclusion Criteria:

* Individuals with developmental disabilities such as mental retardation, autism, and Down syndrome, severe cognitive limitations following stroke, or diagnoses of severe psychopathology will be excluded from participation as these disorders have the potential to confound the findings.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population are youths with sickle cell disease who are experiencing intermittent pain episodes that interfere with quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B McClellan, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- Children's Cancer and Blood Disorder, Columbia, South Carolina, United States

REFERENCES:
- [Background] McClellan CB, Schatz JC, Puffer E, Sanchez CE, Stancil MT, Roberts CW. Use of handheld wireless technology for a home-based sickle cell pain management protocol. J Pediatr Psychol. 2009 Jun;34(5):564-73. doi: 10.1093/jpepsy/jsn121. Epub 2008 Nov 23. PMID 19029141
- [Derived] Schatz J, Schlenz AM, McClellan CB, Puffer ES, Hardy S, Pfeiffer M, Roberts CW. Changes in coping, pain, and activity after cognitive-behavioral training: a randomized clinical trial for pediatric sickle cell disease using smartphones. Clin J Pain. 2015 Jun;31(6):536-47. doi: 10.1097/AJP.0000000000000183. PMID 25503599